CLINICAL TRIAL: NCT02630225
Title: Helping Individuals With Firearm Injuries: A Cluster Randomized Trial
Brief Title: Helping Individuals With Firearm Injuries
Acronym: HIFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency); City of Seattle (Unknown); Arnold Ventures (Unknown)
Responsible Party: Principal Investigator, Ali Rowhani-Rahbar, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000852
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Wounds, Gunshot
Keywords: case management; motivational interviewing
MeSH Terms: conditions — Wounds, Gunshot | interventions — Therapeutics; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive three intervention services in addition to treatment as usual services:
  1. A brief intervention including a feedback session utilizing principles of Motivational Interviewing (MI).
  2. Extended outreach services (6 months) using the Critical Time Intervention (CTI) approach.
  3. Multi-agency attention.
  Interventions: Behavioral: Critical Time Intervention; Other: Treatment as Usual; Behavioral: Motivational Interviewing; Other: Multi-Agency Attention
- Treatment as Usual (Other): Participants in this arm will receive the usual care offered to victims of gun shot wounds.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Critical Time Intervention — The Critical Time Intervention approach strengthens an individual's long-term ties to services, family and friends as well as provides emotional and practical support to individuals during the critical time of transition back to the community. CTI contains three phases:
  Phase 1 - The Support Specialist gets to know the individual, assesses the individual's need and implements a transition plan intended to link the individual to services and supports in the community.
  Phase 2 -- The Support Specialist monitors and adjusts the systems of support that were developed in Phase 1.
  Phase 3 -- The Support Specialist helps the individual develop and implement a plan to achieve long-term goals and finalizes the transfer of responsibilities to caregivers and community providers.
  Arms: Intervention
Other: Treatment as Usual — Services provided by HMC physicians and staff that are part of standard care for patients with firearm-related injuries. This care could include:
  1. All necessary medical care and scheduled follow-ups with subspecialty services
  2. Evaluation by social work with referral to appropriate community services
  3. Screening for alcohol use
  4. Discharge planning services
  5. Financial counseling
Behavioral: Motivational Interviewing — A brief intervention to elicit the goals and needs of participants. As needed, this will included referrals to community resources.
  Arms: Intervention
Other: Multi-Agency Attention — Intervention cases will receive attention from a multidisciplinary team of professionals. This team will help the study Support Specialist identify service recommendations and provide case management guidance.
  Arms: Intervention

SUMMARY:
The investigators will conduct a cluster randomized trial of an intervention program that combines a hospital-based intervention, structured outreach program, and multi-agency attention. The goal of the study is to test the effect of this multi-component intervention on criminal activity, injury, substance abuse, mental health, quality of life, violent behavior, and death.

Investigators aim to enroll a total of 300 patients admitted to the Harborview Medical Center (HMC) for firearm-related injuries. Patients will be randomized to receive a multi-component intervention or treatment as usual. All participants will complete surveys at the time of study consent (baseline) and then at designated time points for 12 months post-consent. Study staff will routinely collect participant records from Washington State Patrol records, HMC medical records, Washington State trauma registry, Washington State Emergency Department Information Exchange, Administrative Office of the Courts, and vital records. The investigators will test the impact of the intervention against standard care. The hypothesis is that participants in the intervention group will see greater improvements in aforementioned outcomes than those in the control group.

DETAILED DESCRIPTION:
About 250 individuals present to an emergency department in King County, primarily Harborview Medical Center (HMC), for firearm-related injuries each year. Almost two-third of these patients require admission for their injuries. While the number of patients with firearm injuries who present to HMC is relatively small, these individuals are at substantially increased risk of subsequent re-hospitalization for another firearm or assault-related injury, arrest for firearm-related or violent crime, non-firearm-related nonviolent crime or firearm-related death in the five years after discharge from the hospital. Thus, interventions among this high risk population have the potential to reduce recidivism, morbidity, and mortality as well as decrease firearm violence and its consequences in the community.

Patients with gunshot wounds (GSWs) seen at HMC receive many services; however, currently there is no standardized intervention offered to GSW patients. A number of hospitals across the country have created violence prevention and intervention programs to help patients who sustain violent injuries. These programs engage patients in the hospital during their recovery period, which is seen as an opportunity ("teachable moment") to change their life and reduce retaliation and recidivism. As a result of the growing number of violence prevention and intervention program, the National Network of Hospital-based Violence Intervention Programs, has been established. Through working groups, meetings, e-newsletter, and conferences, Network members collaborate in research and evaluation, explore opportunities for funding sustainability, develop and share best practices, and identify ways to collectively have an impact on policy. While the creation of this infrastructure is a step in the right direction, researchers have not rigorously tested the effectiveness of these intervention programs. Specifically, no trials have evaluated the effectiveness of hospital-based violence intervention programs offered to GSW victims.

The investigators aim to conduct a cluster randomized trial of an violence intervention program that combines a brief, hospital-based intervention, a structured outreach program, and multi-agency attention. Study staff will provide a brief intervention derived from motivational interviewing (MI). MI is is a patient-centered behavioral technique based on the stages of change model and attempts to engage patients in order to find reason to change behavior. By empathetically exploring ambivalent feelings about health-related behavior, MI encourages reduction in risky behavior. Research has demonstrated the effectiveness of providing MI-based brief interventions in the Emergency Department (ED) or inpatient wards, primarily for alcohol use disorders but also for violent behaviors. Specifically, brief, MI interventions have been successful at reducing youth violence in large urban populations, with effects sustained through one year. Additionally, a behavioral-based intervention including MI targeting adolescents admitted to HMC with trauma showed a reduction in weapon carriage during the year post-hospitalization.

A longitudinal outreach intervention program provides the added benefit of continued engagement. GSW patients must transition back to the community after their hospitalization, and the transitional period, when patients must navigate a complex and fragmented system of care, is especially challenging. Providing GSW patients with outreach and follow-up after the healthcare encounter holds promise for reducing their future violence and criminal activity. The Critical Time Intervention (CTI) approach may provide a strong framework for providing these patients with appropriate outreach and follow-up. Strong evidence supports CTI's effectiveness. The CTI model meets the Coalition for Evidence-based Policy's rigorous "Top Tier" standard for interventions: well-designed and implemented randomized controlled trials, preferably conducted in typical community settings, [that] produced sizable, sustained benefits to participants and/or society. CTI is a time-limited, evidence-based case management model that mobilizes support for society's most vulnerable individuals during periods of transition such as discharge from inpatient services to the community. It facilitates community integration and continuity of care by ensuring that a person has enduring ties to their community and support systems during these critical periods. CTI has been used worldwide among veterans, people with mental illness, homeless or incarcerated individuals, and many other groups. From the beginning, CTI was thought of as an intervention that could be applied in myriad contexts. This approach has the potential to provide an intervention framework for a second tier outreach to GSW victims in King and neighboring counties.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent within 4 weeks following hospital discharge
* Able to understand and speak English
* Able to provide at least one mode of direct or alternate contact (e.g., cell phone, land line, e-mail, friend, or relative)
* Planning to live in King, Pierce, Snohomish, Thurston or Yakima counties for at least 6 months subsequent to hospital discharge
* Receiving treatment for a GSW at HMC and returning to the community, and not prison following treatment
* Being treated for gunshot wounds from assaults or accidents (self- or other-inflicted)

Exclusion Criteria:

* 17 years of age or younger
* Unable to provide consent (including those with severe neurologic damage) within 4 weeks following hospital discharge
* Unable to understand or speak English
* Unable to provide any mode of direct or alternate contact
* Not living in King, Pierce, Snohomish, Thurston or Yakima counties, or planning to move outside of those counties within 6 months following hospital discharge
* Not receiving treatment for a GSW at HMC
* Not returning to the community following hospital discharge (e.g., being sent to a rehabilitation center, skilled nursing facility, or prison)
* Incarcerated at the time of GSW injury
* Being treated for an intentional, self-inflicted gunshot wound injuries (e.g. suicide attempts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Criminal Activity - Records | Two years
  Criminal activity will be measured using Washington State arrest reports and charges from the Administrative Office of the Courts for any violent or nonviolent crime

SECONDARY OUTCOMES:
Injury | Two years
  Injury will be measured using information from medical records, the Washington State Comprehensive Hospital Abstract Reporting System, and the Emergency Department Information Exchange.
Death | Two years
  All cause and cause-specific mortality will be measured using vital records.
Impulsive-Premeditated Aggression Behavior | One year
  This behavior will be measured using the Impulsive-Premeditated Aggression Scale (IPAS).
Interpersonal Violence | One year
  Interpersonal violence will be measured using Conflict Tactics Scale.
Alcohol Use | One year
  Alcohol use will be measured using the the Alcohol Use Identification Test (AUDIT).
Drug Abuse | One year
  Drug abuse will be measured using The National Institute on Drug Abuse - Modified Alcohol, Smoking and Substance Abuse Involvement Screening Test (NIDA - Modified ASSIST).
Posttraumatic Stress Disorder (PTSD) | One year
  PTSD will be measured using the Posttraumatic Stress Disorder (PTSD) Checklist - Civilian Version (PCL-C).
Depression | One year
  Depression will be measured using the Patient Health Questionnaire-8 (PHQ-8).
Employment Status | One year
  This will be measured using survey questions that elicit information about new, continued or discontinued employment.
Educational Attainment | One year
  Education will be measured using survey that elicit information about enrollment in, completion of or discontinuation of educational activities.
Health-Related Quality of Life | One year
  This will be measured using the Short Form Health Survey (SF-12).
Satisfaction with Areas of Life | One year
  Satisfaction with specific areas of life, including study participation, will be measured using the Happiness Scale.
Perceived Social Support | One year
  This will be measured using the Multidimensional Scale of Perceived Social Support.
Housing Status | One year
  Housing status will be measured using survey questions that elicit information about housing circumstances.
Physical and Mental Health Service Utilization | One year
  This will be measured using survey questions that elicit information about use of physical and mental health services.
Criminal Activity - Records | Two years
  Criminal activity will be measured using Washington State arrest reports and charges from the Administrative Office of the Courts differentiating arrests for violent or non-violent crimes.
Criminal Activity - Self Report | One year
  Criminal activity will be measured self-reports of delinquency and criminal activity based on the scale used in the Pittsburgh Youth Study.
Hospitalization - Records | Two years
  Hospitalization will be measured using Washington State Comprehensive Hospital Abstract Reporting System (CHARS)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rowhani-Rahbar, MD, MPH, Principal Investigator — University of Washignton
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Floyd AS, Lyons VH, Whiteside LK, Haggerty KP, Rivara FP, Rowhani-Rahbar A. Barriers to recruitment, retention and intervention delivery in a randomized trial among patients with firearm injuries. Inj Epidemiol. 2021 Jul 26;8(1):37. doi: 10.1186/s40621-021-00331-z. PMID 34304738
- [Derived] Lyons VH, Floyd AS, Griffin E, Wang J, Hajat A, Carone M, Benkeser D, Whiteside LK, Haggerty KP, Rivara FP, Rowhani-Rahbar A. Helping individuals with firearm injuries: A cluster randomized trial. J Trauma Acute Care Surg. 2021 Apr 1;90(4):722-730. doi: 10.1097/TA.0000000000003056. PMID 33405475